CLINICAL TRIAL: NCT05547503
Title: A Double-blind, Placebo-controlled, Study of the Safety, Tolerability, and Pharmacokinetics of Single Ascending Doses of Oral AFA-281 (Phase I Part 1) and Multiple Ascending Doses of Oral AFA-281 (Phase I Part 2) in Healthy Volunteers
Brief Title: Phase I Single Ascending Dose and Multiple Ascending Doses of Oral AFA-281 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Afasci Inc (Industry)
Collaborators: Cognitive Research Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AFA-281-001
Record Dates: First submitted 2022-09-14; First posted 2022-09-21 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Pain, Neuropathic; Pain, Inflammatory
MeSH Terms: conditions — Neuralgia; Pain

STUDY DESIGN:
Intervention Model Description: Part 1: Single escalation dose Part 2: Multiple escalation doses for 14 days
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Part 1 and Part 2 studies are double-blind placebo controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo Control (Placebo Comparator): Double blind placebo control
  Interventions: Drug: AFA-281
- AFA-281 (Experimental): Part 1: AFA-281 administered as an oral capsule at 5 dose levels for one day.
  Part 2: AFA-281 administered as an oral capsule at 3 dose levels twice daily for 14 consecutive days. Doses will be determined after completion of Part 1.
  Interventions: Drug: AFA-281

INTERVENTIONS:
Drug: AFA-281 — Part 1: AFA-281 will be administered as a single dose at 4 dose levels (TBD) Part 2: AFA-281 will be administered twice daily for 14 - 21 days at 3 dose levels (TBD)

SUMMARY:
Phase I Part 1 (single ascending dose):

Double-blind dosing will occur in healthy volunteers in 4 cohorts of 8 subjects each. Six subjects in each cohort will be randomized to receive AFA-281 and 2 subjects will be randomized to receive the matching placebo. At the end of the Part 1 study is to evaluate the safety and tolerability of AFA-281. Following completion of each cohort, bioanalytical analyses will be conducted to evaluate the pharmacokinetic profile.

Phase I Part 2 (multiple dose for 14 days):

Pending the results from Part 1, healthy volunteers will be administered AFA-281 for 14 to 21 consecutive days in 3 cohorts. At scheduled intervals after dosing, and at the end of the cohort's study period to evaluate the safety and tolerability and the pharmacokinetic profile of AFA-281.

DETAILED DESCRIPTION:
Phase I Part 1 (single ascending dose):

Healthy volunteers will be admitted to the clinical research unit on Day -1. There will be five cohorts with 8 subjects per cohort. Six subjects per cohort will receive AFA-281 at one of 4 doses and 2 will receive placebo. Oral capsules will be administered on the morning of Day 1, following a 10-hour fast. Blood draws for assessment of Pharmacokinetic parameters will occur 0.2-1 hr pre-dose and at 0.5-, 1-, 2-, 3-, 4-, 8-, 10, 12-, 16-, 24-, 36-, 48-hr, and up to 72-hr post-dose. Vital signs will be collected at scheduled times following dosing. A 12-lead ECG will be obtained pre-dose and scheduled at 2, 4, 8, 24 hr, and 3- or 4 days post- dose. Various clinical laboratory tests will be drawn on Day -1, within 1 hr prior to dosing, and at scheduled timepoints after dosing while the volunteer is housed in the research center. Subjects of Cohorts 1 - 3 will be released following completion of blood draws and safety assessments up to 48 hours and Cohorts 4 and 5 subjects will return for 72-hour blood draws and Day 4 ECG and safety assessment.

Phase I Part 2 (multiple ascending doses - 14 days):

After assessment of the safety data from the single dose Phase I Part 1, healthy volunteers will be randomized into 3 cohorts with 8 subjects per cohort. Five subjects per cohort will receive AFA-281 and 3 will receive placebo. Oral capsules will be administered in dose titration and split daily dose in fours time daily (QID) for 14 - 21 consecutive days. Routine clinical monitoring will occur as in Part 1. Baseline physical examination, vital signs, clinical lab tests, and ECGs will be performed prior to dosing, at scheduled intervals after dosing, and at the end of the cohort's study period to evaluate the safety and tolerability, and the pharmacokinetic profile of AFA-281. Reports of potential adverse events will be elicited, and vital signs and 12-lead ECG will be measured in a similar manner to Part 1. Similarly, clinical laboratory tests will be drawn prior to and after dosing.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be in good general health with no significant medical history and have no clinically significant abnormalities on physical examination at screening and/or before administration of the initial dose of study drug.

  * Participants must have a Body Mass Index (BMI) between 18.0 and 30.0 kg/m2 inclusive.
  * Participants must have clinical laboratory values within normal range as specified by the testing laboratory, unless deemed not clinically significant by the Investigator or delegate.
  * Participants must have an ECG without clinically significant pathologic abnormalities.

Exclusion Criteria:

* Participants with significant medical history or clinically significant abnormalities
* Participants with clinically significantly pathologic abnormalities
* Participants with ECG abnormalities

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2023-04-11 (Actual); Primary Completion 2024-12-04 (Actual); Study Completion 2025-05-14 (Actual)

PRIMARY OUTCOMES:
Treatment-Related Adverse Events | Predose and Up to 72 hours after dose
  Number of participants with treatment-related adverse events will be assessed using CTCAE v5.0
Heart rate | Predose and Up to 72 hours after dose
  Heart rate as one of vital signs will be measured
Body temperature | Predose and Up to 72 hours after dose
  Body temperature (0C) as one of vital signs will be measured
Blood Pressure | Predose and Up to 72 hours after dose
  Blood pressure as one of vital signs will be measured
Electrocardiogram (ECG) | Pre-dose and up to 72 hours after dose
  Triplicate 12-lead ECG will be measured to evaluate electrical activity of the heart
Blood chemistry | Pre-dose and up to 72 hours after dose
  Blood chemistry parameters will be measured
Hematology | Pre-dose and up to 72 hours after dose
  Hematology parameters will be measured
Coagulation | Pre-dose and up to 72 hours after dose
  Coagulation parameters (PT/INR, PTT) will be measured
Urinalysis | Pre-dose and up to 72 hours after dose
  Urinalysis parameters will be measured using dipstick and microscopic examination.
Blood maximum plasma concentration (Cmax) of the study drug | Pre-dose and up to 72 hours after dose
  Pharmacokinetics parameter Cmax will be measured to assess drug exposure levels in blood
Blood study drug half-life (t1/2) | Pre-dose and up to 72 hours after dose
  Pharmacokinetics parameter t1/2 will be measured to evaluate drug half-life in the blood
Area under the plasma concentration versus time curve (AUC) of the study drug | Pre-dose and up to 72 hours after dose
  Pharmacokinetics parameter AUC will be measured

SECONDARY OUTCOMES:
A dose and exposure relationship | Pre-dose and up to 72 hours after dose
  Doses of study drug and blood exposure levels will be analyzed to determine dose proportionality.
Tmax of the study drug (parent compound) in blood | Up to 72 hours after dose
  Pharmacokinetics parameter Time at which Cmax of the study drug appeared will be determined.
Plasma Concentration (Cmax) of the major metabolite in blood | Up to 72 hours after dose
  Pharmacokinetics parameter Cmax of a major metabolite will be measured.
Area under the plasma concentration versus time curve (AUC) of the major metabolite in blood | Up to 72 hours after dose
  Pharmacokinetics parameter AUC of a major metabolite will be measured.
The major metabolite half-life (t1/2) in blood | Up to 72 hours after dose
  Pharmacokinetics parameter t1/2 of a major metabolite will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Xinmin Xie, MD, PhD, Study Chair — Afasci Inc
Locations (1):
- CenExcel CNS, Los Alamitos, California, United States

IPD SHARING:
Plan to Share IPD: Yes
One year after completion of the study and 6 months after publication
Supporting Information: SAP, ICF
Time Frame: One year after completion of the study and 6 months after publication
Access Criteria: To be added